CLINICAL TRIAL: NCT01194440
Title: A Phase II Prospective Pilot Study Evaluating Efficacy of Intravenous Zoledronic Acid Prophylaxis for Prevention of Aromatase Inhibitor Associated Musculoskeletal Symptoms: ZAP-AIMSS Trial
Brief Title: Zoledronic Acid in Aromatase Inhibitor Induced Musculoskeletal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: J1022; SKCCC J1022 (Other: SKCCC)
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Ductal Carcinoma in Situ; Estrogen Receptor-positive Breast Cancer; Progesterone Receptor-positive Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Letrozole; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I - IV Zoledronic Acid Prophylaxis (Experimental): Patients receive zoledronic acid IV at months 1 and 6. Beginning 14 days after first zoledronic acid infusion, patients receive oral letrozole once daily for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: letrozole; Drug: zoledronic acid

INTERVENTIONS:
Drug: letrozole — Given orally
  Other Names: CGS 20267; Femara; LTZ
Drug: zoledronic acid — Given IV
  Other Names: CGP 42446; CGP42446A; NDC-zoledronate; ZOL 446; zoledronate; Zometa

SUMMARY:
RATIONALE: Zoledronic acid may prevent bone loss and help prevent or lessen musculoskeletal symptoms in women receiving hormone therapy for breast cancer.

PURPOSE: This phase II trial is studying how well zoledronic acid works in preventing musculoskeletal symptoms in post-menopausal women with stage I, stage II, or stage III breast cancer receiving letrozole.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Percentage of women experiencing aromatase inhibitor associated musculoskeletal symptoms (AIMSS) at 1, 3, 6, and 12 months after bisphosphonate therapy, as compared to historical controls.

II. Change in Health Assessment Questionnaire Disability Index (HAQ-DI) score and 1, 3, 6 and 12 months, from baseline, among those receiving bisphosphonate, as compared to historical controls.

SECONDARY OBJECTIVES:

I. Change in pain scores on visual analog scale (VAS) at 1, 3, 6 and 12 months, from baseline, compared to historical controls.

II. Change in amount and/or frequency of oral analgesic use at 1, 3, 6 and 12 months from baseline among those receiving bisphosphonate therapy, as compared to historical controls.

III. Number of patients who discontinue or change aromatase inhibitor (AI) therapy.

IV. Change in menopausal symptoms (NSABP-revised), hot flash frequency (HFRDIS),sleep quality (PSQI), depression score (CESD) and overall quality of life (EuroQOL) in patients at 1, 3, 6 and 12 months from baseline, among those receiving bisphosphonate therapy, as compared to historical controls.

V. Changes in plasma estrogen concentrations at 1, 3, 6 and 12 months from baseline, among those receiving bisphosphonate therapy, as compared to historical controls.

VI. Change in bone mineral density (DEXA scan) at 12 months from baseline, among those receiving bisphosphonate therapy, as compared to historical controls.

VII. Change in bone turn over markers (serum-C telopeptide, bone-specific alkaline phosphatase, osteocalcin and urinary N-telopeptide) at 1, 3, 6 and 12 months from baseline, among those receiving bisphosphonate therapy, as compared to historical controls.

VIII. Change in inflammatory markers (ESR, CRP, IL-1, IL-6, IL-8) at 1, 3, 6 and 12 months from baseline, among those receiving bisphosphonate therapy, as compared to historical controls.

OUTLINE: Patients receive zoledronic acid intravenously (IV) at months 1 and 6. Beginning 14 days after first zoledronic acid infusion, patients receive oral letrozole once daily for 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria

* Patients with histologically proven DCIS or stage I-III invasive carcinoma of the breast that is estrogen and/or progesterone receptor positive by immunohistochemical staining who are considering aromatase inhibitor therapy; women may receive the AI on this study as initial adjuvant hormonal treatment or following tamoxifen; patients must have completed any adjuvant chemotherapy; patients may have received preoperative chemotherapy
* Postmenopausal status, defined as: >= 60 years of age; or < 60 years of age and amenorrheic for >= 12 months prior to day 1 if intact uterus/ovaries; or < 60 years of age, and the last menstrual period 6-12 months prior to day 1, if intact uterus/ovaries and meets biochemical criteria for menopause (FSH and estradiol within institutional standards for postmenopausal status); or < 60 years of age, without a uterus, and meets biochemical criteria for menopause (FSH and estradiol within institutional standards for postmenopausal status); or < 60 years of age and history of bilateral oophorectomy; or prior radiation castration with amenorrhea for at least 6 months; < 60 years of age and taking medication designed to suppress ovarian function and meets biochemical criteria for menopause (estradiol levels within institutional standards for postmenopausal status; women would have had to be taking the drug for at least 30 days prior to day 1)
* ECOG performance status 0-2
* Patient is aware of the nature of her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form

Exclusion Criteria

* Concurrent use of hormone replacement therapy
* Concurrent use of tamoxifen; patients taking tamoxifen must discontinue the drug prior to first dose of zoledronic acid
* Concurrent use of other selective estrogen receptor modulator (SERM) such as raloxifene
* Concurrent consumption of soy supplements; routine dietary consumption of soy containing foods will be permitted
* Prior use of an aromatase inhibitor in any setting
* Current bisphosphonate use (oral or intravenous); prior bisphosphonate users would be eligible as long as the use was > 1 month ago for oral bisphosphonates and/or > 12 months ago for intravenous bisphosphonates, prior to starting study treatment
* Moderate to severe renal impairment (serum creatinine greater than 2 mg/dL or creatinine clearance less than 50 mL/min)
* Hypersensitivity to letrozole or zoledronic acid or any of its excipients
* Concomitant treatment with oral or intravenous corticosteroids
* Current active dental problems including infection or the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2011 to January 2013, 59 women signed consent, met eligibility criteria, and received study intervention on this clinical trial at the Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins.
Pre-assignment Details: 3 participants were screen failures and 1 participant withdrew consent prior to assignment to treatment.
Groups:
- Arm I - IV Zoledronic Acid Prophylaxis: Patients receive zoledronic acid IV at months 1 and 6. Beginning 14 days after first zoledronic acid infusion, patients receive oral letrozole once daily for 12 months in the absence of disease progression or unacceptable toxicity.
  letrozole: Given orally
  zoledronic acid: Given IV
  laboratory biomarker analysis: Correlative studies
  enzyme-linked immunosorbent assay: Correlative studies
  mass spectrometry: Correlative studies
  bone scan: Correlative studies
  quality-of-life assessment: Ancillary studies
  questionnaire administration: Ancillary studies
  pharmacogenomic studies: Correlative studies
  high performance liquid chromatography: Correlative studies
Period: Baseline (First Dose)
Arm/Group | Arm I - IV Zoledronic Acid Prophylaxis
Started | 59
Completed | 52
Not Completed | 7
Not completed — Reason not specified | 4
Not completed — Lack of Efficacy | 1
Not completed — Change in therapy | 1
Not completed — Adverse Event | 1
Period: 6-months (2nd Dose)
Arm/Group | Arm I - IV Zoledronic Acid Prophylaxis
Started | 52
Completed | 48
Not Completed | 4
Not completed — Change in therapy | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive zoledronic acid IV at months 1 and 6. Beginning 14 days after first zoledronic acid infusion, patients receive oral letrozole once daily for 12 months in the absence of disease progression or unacceptable toxicity.
  letrozole: Given orally
  zoledronic acid: Given IV
  laboratory biomarker analysis: Correlative studies
  enzyme-linked immunosorbent assay: Correlative studies
  mass spectrometry: Correlative studies
  bone scan: Correlative studies
  quality-of-life assessment: Ancillary studies
  questionnaire administration: Ancillary studies
  pharmacogenomic studies: Correlative studies
  high performance liquid chromatography: Correlative studies
Arm/Group | Arm I
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 59
Participants | 22
Statistical Analysis 1: Comparison: Arm I; The primary hypothesis of the study is that administration of zoledronic acid with letrozole would result in a significant decline in the percentage of women experiencing AIMSS compared to letrozole treatment alone (historical control); Test type: Superiority or Other; p < 0.001, Bonferonni; Adjusting for multiple comparisons in the analyses, a Bonferonni-corrected p-value of 0.05/5 = 0.01 to represent statistical significance was used

2. Secondary Outcome: AIMSS as Determined by Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The HAQ-DI score ranges from 0-3 with a higher score reflective of greater disability or increased incidence of AIMSS.
Time Frame: Baseline, 1 month, 3 months, 6 months, 12 months
Population: Data was only collected in 58 participants at baseline, 52 participants at 1 month, 56 participants at 3 months, 51 participants at 6 months, and 45 participants at 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I
Number analyzed (Participants) | 58
score on a scale
  Baseline | 0.2 [0.1 to 0.9]
  1 month: number analyzed (Participants) | 52
  1 month | 0.2 [0.1 to 1.1]
  3 months: number analyzed (Participants) | 56
  3 months | 0.1 [0.1 to 1.2]
  6 months: number analyzed (Participants) | 51
  6 months | 0.2 [0.1 to 1.1]
  12 months: number analyzed (Participants) | 45
  12 months | 0.4 [0.1 to 2.2]

3. Secondary Outcome: AIMSS as Determined by Visual Analog Scale (VAS) Score
Description: VAS is a visual measurement tool to assess AIMSS. It is a visual scale that ranges from 0 centimeters (cm) to 10cm. The VAS score ranges from zero (0cm) to 10 (10cm), with a higher score reflecting a greater frequency of AIMSS.
Time Frame: Baseline, 1 month, 3 months, 6 months, 12 months
Population: Data was only collected for 58 participants at baseline, 52 participants at 1 month, 55 participants at 3 months, 50 participants at 6 months, and 45 participants at 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I - IV Zoledronic Acid Prophylaxis
Number analyzed (Participants) | 58
score on a scale
  Baseline | 0.8 [0 to 8.3]
  1 month: number analyzed (Participants) | 52
  1 month | 1 [0.1 to 8.1]
  3 months: number analyzed (Participants) | 55
  3 months | 1.4 [0.2 to 8.8]
  6 months: number analyzed (Participants) | 50
  6 months | 1.2 [0.1 to 7]
  12 months: number analyzed (Participants) | 45
  12 months | 1.9 [0.1 to 9.7]

4. Secondary Outcome: Number of Participants Who Discontinue or Change Aromatase Inhibitor (AI) Therapy
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 59
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 12 month intervention period.
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 53/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=59)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Chills (General disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Edema Limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 12 (12)
Fever (General disorders) | 6 (6)
Flu-Like Symptoms (General disorders) | 9 (9)
Hot Flashes (Vascular disorders) | 36 (36)
Insomnia (Psychiatric disorders) | 11 (11)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 11 (11)
Memory Impairment (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7)
Neuralgia (Nervous system disorders) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 16 (16)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (4)
Vaginal Dryness (Reproductive system and breast disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes